CLINICAL TRIAL: NCT07365722
Title: Minimally-Invasive Non-Surgical Therapy Of Peri-implantitis: A Multicenter Randomized Controlled Trial
Brief Title: Comparison of Two Non-surgical Procedure to Manage Gum Disease Around Implants.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 51376
Record Dates: First submitted 2026-01-05; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Peri Implantitis
Keywords: peri implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomisation lists for each centre will be generated by an independent researcher, who will be involved in the study. The examiners, who assess the clinical variables, will be blinded with regards to the patients' treatment assignments. The measures will include no access to the dental records as to which treatment has been assigned and no access to the patients' treatment file.
  The statistician who will perform the statistical analyses, will have no access to the allocation of the patients into the respective treatment group.
  The clinician cannot be blinded since she/he has to handle the different devices, but she/he will have no access to the data collection sheets or the group allocation. The assistant to the clinician cannot be blinded since she/he has to handle the different devices, but she/he will have no access to the data collection sheets or the group allocation. The patients will be not blinded to the treatment provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Surgical Periodontal Therapy- Group (Active Comparator): Control group will receive one session of non-surgical debridement as described previously (Liñares et al., 2019) by an experienced periodontist. Non-surgical treatment under local anaesthesia consisting of supra- and submucosal mechanical debridement using ultrasonic stainless steel scaling inserts(EMS® , Electro Medical Systems) will be performed in one treatment session with no time restrictions. After that, a stainless steel Columbia 4R/4L curette (LM Instruments Oy) will be used to remove granulation tissue and minor mucosal curettage.
  Interventions: Procedure: Non-Surgical Periodontal treatment (NSPT)
- Minimally-invasive non-surgical therapy of peri-implantitis- Group (Experimental): Minimally-invasive non-surgical therapy of peri-implantitis
  Half of the study participants (tests) will be randomised to receive minimally-invasive non-surgical periodontal treatment (MINST). All treatment will be carried out by the same therapist in each centre, including oral hygiene. The protocol for MINST is as follows: participants will receive local anaesthesia, then thorough debridement of the implant surface will be completed to the depth of the periodontal and peri-implant pockets following this protocol:
  * In agreement with (Mehta et al., 2024) exclusive use of piezo-electric/ultrasonic devices with specific non-diamond thin and delicate tips (PS, PL1, PL2 from EMS, Nyon, Switzerland; Siroperio 1, 2, 3 and 7 from Sirona, Salzburg, Austria; Woodpecker P3 tip, Guilin Woodpecker, Guilin, China; Satelec 10Z from Acteon, UK, depending on what was available in the different study centres)
  * using at least x3 magnification loupes
  * aiming to obtain a stable blood clot in the pock
  Interventions: Procedure: Minimally-invasive non-surgical therapy of peri-implantitis

INTERVENTIONS:
Procedure: Non-Surgical Periodontal treatment (NSPT) — Control group will receive one session of non-surgical debridement as described previously (Liñares et al., 2019) by an experienced periodontist. Non-surgical treatment under local anaesthesia consisting of supra- and submucosal mechanical debridement using ultrasonic stainless steel scaling inserts(EMS® , Electro Medical Systems) will be performed in one treatment session with no time restrictions. After that, a stainless steel Columbia 4R/4L curette (LM Instruments Oy) will be used to remove granulation tissue and minor mucosal curettage.
  Arms: Non Surgical Periodontal Therapy- Group
Procedure: Minimally-invasive non-surgical therapy of peri-implantitis — Half of the study participants (tests) will be randomised to receive minimally-invasive non-surgical periodontal treatment (MINST). All treatment will be carried out by the same therapist in each centre, including oral hygiene. The protocol for MINST is as follows: participants will receive local anaesthesia, then thorough debridement of the implant surface will be completed to the depth of the periodontal and peri-implant pockets following this protocol:
  * In agreement with (Mehta et al., 2024) exclusive use of piezo-electric/ultrasonic devices with specific non-diamond thin and delicate tips (PS, PL1, PL2 from EMS, Nyon, Switzerland; Siroperio 1, 2, 3 and 7 from Sirona, Salzburg, Austria; Woodpecker P3 tip, Guilin Woodpecker, Guilin, China; Satelec 10Z from Acteon, UK, depending on what was available in the different study centres)
  * using at least x3 magnification loupes
  * aiming to obtain a stable blood clot in the pocke
  Arms: Minimally-invasive non-surgical therapy of peri-implantitis- Group

SUMMARY:
Research Question:

Can a minimally invasive, non-surgical treatment approach (MINST) be more effective than the current standard non-surgical method in treating peri-implantitis, a common inflammatory condition affecting dental implants?

Background:

Dental implants are widely used to replace missing teeth. While they are usually successful, some patients develop a condition called peri-implantitis, an infection that causes inflammation and bone loss around the implant. This can eventually lead to implant failure if not treated properly. Currently, non-surgical treatments are used to clean the area and reduce inflammation. However, these methods often fall short of fully resolving the issue, and many patients require further treatment or even surgery.

A newer approach called MINST (Minimally-Invasive Non-Surgical Therapy) has shown promising results for treating gum disease around natural teeth. This method focuses on precision cleaning with minimal trauma to the surrounding tissues, reducing pain and improving healing. While MINST works well for gum disease, its effectiveness for treating peri-implantitis has not yet been tested.

Purpose of the Study:

This clinical trial will compare the effectiveness of MINST with the standard non-surgical treatment currently used for peri-implantitis.

The aim is to determine whether MINST can better treat the disease, improve healing, and reduce discomfort for patients.

Hypotheses:

Alternate Hypothesis (What we expect to find): MINST will result in better outcomes, specifically, fewer deep pockets around the implant, less bleeding, and fewer signs of infection, compared to the standard treatment.

Null Hypothesis: There will be no significant difference between the outcomes of the two treatment approaches.

Study Design:

Type of Study: A randomized controlled trial (RCT) involving 106 patients. Duration: Patients will be followed for 12 months after treatment. Locations: Multiple dental centers participating in the trial. Method: Half of the participants will receive MINST; the other half will receive the standard treatment. Neither patients nor outcome assessors will know which treatment was used (single-masked). What Will Be Measured? Primary Goal: To see how many patients show healing (defined as smaller pockets, little or no bleeding, and no pus) 12 months after treatment.

Secondary Goals:

Patient-reported outcomes, including pain levels and quality of life Changes in pocket depth and tissue attachment Bacterial changes Time taken for treatment appointments Why Is This Important? If MINST proves to be more effective and comfortable for patients, it could change how peri-implantitis is managed in the future- potentially reducing the need for surgery, improving patient experience, and helping more people keep their dental implants for longer.

DETAILED DESCRIPTION:
Study Overview (Design) This is a research study being carried out at several dental clinics to test two different types of non-surgical treatments for periimplantitis- a condition where the tissues around a dental implant become infected and inflamed. The goal is to see which treatment works better over a period of 12 months. Study Schedule Participants will be followed for 1 year after their treatment, with several check-up visits to monitor progress and collect information.

Who Can Take Part? Inclusion (Who can join?) People with peri-implantitis, a condition affecting the gums and bone around a dental implant.

At least one area around the implant with deep pockets (>6mm) and some bone loss.

Page 8 of 23 Project ID: 51376 Implants must be accessible for cleaning without removing the crown or prosthetic.

Good general mouth hygiene (low plaque and bleeding scores). Exclusion (Who cannot join?) People who recently took antibiotics. Pregnant or breastfeeding women. Those with certain medical conditions (e.g., uncontrolled diabetes). People who already had treatment for this condition recently. Smokers or people who vape. Implants that are severely damaged or considered untreatable. Recruiting Patients Patients referred to specialist periodontal clinics will be checked to see if they qualify. If they do, they'll be informed about the study and can decide whether to participate. If they agree, they will attend a baseline appointment where their current oral health will be recorded. Randomisation (Choosing Treatment Groups)

Participants will be randomly assigned to one of two treatment groups:

Standard non-surgical treatment Minimally invasive non-surgical treatment (MINST) The method of choosing who goes into which group is like flipping a coin-but controlled by a secure computer system to ensure fairness. Blinding/Masking (Avoiding Bias) The dentist doing the treatment will know which method is being used (they have to, to apply the treatment correctly).

But the person who checks the results (examiner) and the person analyzing the data (statistician) won't know who received which treatment. This helps make the study results more reliable. Patients will know which treatment they received. Treatment and Follow-up Visits

Participants will attend up to 7 visits over 12 months:

Visit 1 (Day 0 - Baseline) Consent to take part Full dental and medical check Photos taken Oral hygiene advice Visit 2 (Treatment)

One of the two types of cleaning will be performed:

Standard: Cleaning using ultrasonic tools and curettes. MINST: Cleaning using finer tools and magnification for a more gentle and precise approach.

Visit 3 (1 Month) Follow-up with oral hygiene support Check for pain or discomfort Short cleaning if needed Visit 4 (3 Months) - Optional Check-up with hygiene instructions Visit 5 (6 Months) Page 9 of 23 Project ID: 51376 Full periodontal check Cleaning and photos Visit 6 (9 Months) - Optional Same as 6-month visit Visit 7 (12 Months) Final check-up with full periodontal exam and photos Study completed Rescue Treatment (If Needed)

If the implant doesn't improve or worsens during the study, the patient may receive additional treatment, which could include:

Extra cleaning Surgery In serious cases, implant removal These situations will be documented and analyzed. Clinical Measurements

At various visits, the study team will:

Measure gum pocket depths around teeth and implants. Record bleeding, gum recession, plaque, and other oral health signs. Use a standard dental probe for measurements at six points around each implant and tooth.

Photographs Photos and sometimes videos will be taken to monitor changes over time. These will be stored securely and anonymised to protect patient privacy. PROMs (Patient-Reported Outcomes) Patients will fill in questionnaires at several time points (baseline, 4, 8, and 12 months) to report how their mouth condition affects their daily life. One is a general oral health quality-of-life questionnaire (OHIP-14), and another is implant-specific.

Repeatability (Calibration) To make sure the measurements are accurate and consistent, all examiners will go through training and calibration exercises before the study starts. X-rays Previous X-rays (taken within the last 3 months) will be used to confirm the bone loss around the implant. No new X-rays will be taken solely for the study. End of Study The study ends one year after the last patient finishes their follow-up. After that, patients can choose to be monitored annually for up to 4 more years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peri-implantitis (any implant surface/any amount of keratinized gingiva)
* PPD>6mm at least in one implant surface
* Bone levels ≥3mm apical of the most coronal portion of the intra-osseous part of the implant.
* Implant surface deemed accessible by the treating clinician, without the need to remove the prosthetic suprastructure
* Full-mouth plaque score <30%
* Full-mouth bleeding score <30%

Exclusion Criteria:

* A course of antibiotics within the past 3 months
* Pregnant/lactating women
* Relevant medical history as evaluated by the examining clinician which may have the potential to affect periodontal surgical treatment (e.g., uncontrolled diabetes HbA1c≥7).
* Individuals on long-standing (2 or above years) supportive peri-implant care (SPIC)
* Previous non-surgical or surgical therapy of the affected implant within 12 months
* Current smoking or vaping (defined as any smoking or vaping within 12 months)
* Implant considered hopeless according to the treating clinician (e.g. mobility, circumferential bone loss >80%, implant outside the bone envelope)
* Case needing adjunctive antibiotic therapy, according to the treating clinician

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-02-07 (Estimated)

PRIMARY OUTCOMES:
Probing Pocket depth | 12 months
  measure in mm of distance between gingival margin and bottom of the periodontal pocket

SECONDARY OUTCOMES:
Bleeding on probing | 12 months
  presence or absence of bleeding after probing the periodontal pocket
suppuration | 12 months
  presence or absence of suppuration after probing the periodontal pocket

IPD SHARING:
Plan to Share IPD: Yes
upon requested to the authors
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code